CLINICAL TRIAL: NCT01228084
Title: The Effects of Sulforaphane in Patients With Biochemical Recurrence of Prostate Cancer
Brief Title: Sulforaphane in Treating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: The Wayne D. Kuni and Joan E. Kuni Foundation (Other)
Responsible Party: Principal Investigator, Joshi Alumkal, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6613; SOL-10082-L (Other: OHSU Knight Cancer Institute); 6613 (Other: OHSU IRB)
Record Dates: First submitted 2010-10-19; First posted 2010-10-25 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer
Keywords: sulforaphane; broccoli sprout extract (BSE); prostate cancer; recurrent prostate cancer; phase II
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulforaphane (Experimental): Sulforaphane given 200μmol (total daily) orally in four 50μmol capsules taken once daily from Week 1 Day 1 to Week 20 Day 7. On days when clinic visits are required patient must wait to take that day's dose until instructed to do so in clinic.
  Interventions: Drug: Sulforaphane; Other: Laboratory biomarker analysis; Other: Pharmacological study

INTERVENTIONS:
Drug: Sulforaphane — Sulforaphane given 200μmol (total daily) orally in four 50μmol capsules taken once daily from Week 1 Day 1 to Week 20 Day 7. On days when clinic visits are required patient must wait to take that day's dose until instructed to do so in clinic.
  Other Names: Broccoli Sprout Extract (BSE)
Other: Laboratory biomarker analysis — Correlative studies
Other: Pharmacological study — Correlative studies
  Other Names: Pharmacological studies

SUMMARY:
This phase II trial studies how well sulforaphane works in treating patients with recurrent prostate cancer. Sulforaphane may prevent or slow the growth of certain cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients who achieve a 50% decline in prostate-specific antigen (PSA) levels within 20 weeks of sulforaphane treatment.

SECONDARY OBJECTIVES:

I. To determine the percentage change in PSA from baseline to the final measured value at the end of study as well as the maximal PSA decline that occurs while on study for each subject.

II. To determine the proportion of patients whose PSA has not doubled after full 20 weeks of sulforaphane treatment.

III. To determine the safety profile of sulforaphane. IV. To determine the pharmacokinetics (PK) of sulforaphane and its metabolites in blood.

V. To determine the effect of sulforaphane supplementation on target pharmacodynamic (PD) modulation in peripheral blood cells.

VI. To assess the effect of Glutathione-S-Transferase Mu 1 (GSTM1) genotype on sulforaphane PK, PD.

VII. To collect frozen serum for future analysis of correlative biomarkers.

OUTLINE:

Patients receive sulforaphane orally (PO) once daily for 20 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 14-30 days and every 6 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically proven adenocarcinoma of the prostate treated with either a prostatectomy or definitive radiation (external beam or brachytherapy
* Protocol-Specific Prostate Working Group 2 (PCWG2) Criteria: rising PSA after definitive therapy

  * For post surgical patients: the nadir reference value (#1) is the last PSA measured before increases are documented, with subsequent values obtained a minimum of 1 week apart; if the PSA at time point 3 (value #3A) is greater than that at point 2, then eligibility has been met; if the PSA is not greater than point 2 (value #3B), but value #4 is, the patient is eligible assuming that other criteria are met and values 3A or #4 are 1.0 ng/mL or higher
  * For post radiation therapy patients: the nadir reference value (#1) is the last PSA measured before increases are documented, with subsequent values obtained a minimum of 1 week apart; if the PSA at time point 3 (value #3A) is greater than that at point 2, then eligibility has been met; if the PSA is not greater than point 2 (value #3B), but value #4 is, the patient is eligible assuming that other criteria are met and if values 3A or #4 are 2.0 ng/mL or more above the nadir reference value (#1) according to Phoenix/American Society for Therapeutic Radiology and Oncology (ASTRO) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2
* The following laboratory results within 4 weeks prior to starting study treatment:

  * White blood cells (WBC) >= 3000/mm^3
  * Neutrophil >= 1,500/mm^3
  * Platelet >= 100,000/mm^3
  * Serum creatinine =< upper limit of normal (ULN)
  * Albumin > 3.0 gm/dL
  * Total bilirubin < 1.5 X ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 X ULN
  * Testosterone level >= 150ng/dL, and no evidence of progression while on prior hormonal therapy, if applicable (i.e. patient must be non-castrate resistant).
* Prior androgen therapy is allowed as long as the patient did not progress while on therapy.
* The following imaging scans within 12 weeks prior to starting study treatment: Whole Body Bone Scan: computed tomography (CT) Chest/Abdomen/Pelvis w/ contrast; NOTE: if contrast medium for CT scan is contraindicated for the patient, documentation of this is required and a CT scan with contrast will not be required; subject still must obtain a CT without contrast, though.
* Willingness to use effective contraception by study participants or their female partners throughout the treatment period and for at least 2 months following treatment
* Signed informed patient consent and Health Insurance Portability and Accountability Act (HIPAA) within 3 months prior to starting treatment

Exclusion Criteria:

* Significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* Measurable and/or evaluable recurrent prostate cancer by imaging (CT scan of the chest, abdomen, and pelvis and bone scan performed within 12 weeks prior to starting treatment) or by physical exam
* Prior investigational therapy within 30 days prior to starting study treatment
* Prior treatment with a known histone deacetylase inhibitor (including but not limited to valproic acid, suberoylanilide hydroxamic acid [SAHA],Panobinostat (LBH589), etc) within 6 months prior to starting study treatment or while on study therapy
* Concurrent systemic treatment for prostate cancer
* Current treatment with warfarin
* Gastrointestinal ailments which would interfere with the ability to adequately absorb sulforaphane
* Allergy to cruciferous vegetables
* Any condition which, in the opinion of the study clinician, would make participation in the study harmful to the patient

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshi J Alumkal, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulforaphane
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve a 50% Decline in Prostate-Specific Antigen (PSA) Levels
Description: To determine the proportion of patients who achieve a decline in PSA levels while receiving sulforaphane treatment. as a measure of anti-tumor activity in men with recurrent prostate cancer.
Time Frame: Less than or equal to 20 weeks of sulforaphane treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
percentage of participants | 5

2. Secondary Outcome: Percent Change in PSA From Baseline to Final Measured Value at End of Study
Description: To determine the percentage change in PSA from baseline to the final measured value at the end of study.
Time Frame: Measure at baseline and after stopping study treatment (less than or equal to 20 weeks of treatment with sulforaphane.)
Measure: Median (Full Range); unit: Percent change
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
Percent change | 35 [-32 to 152]

3. Secondary Outcome: Minimum Percent Change in PSA (i.e., the Smallest Increase for Those With Increased PSA and the Greatest Decline for Those With Decreased PSA)
Time Frame: PSA measured every 28 days while on study treatment, an average of 5 months
Measure: Median (Full Range); unit: percent change
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
percent change | 2 [-71 to 48]

4. Secondary Outcome: Proportion of Patients Whose PSA Levels Have Not Doubled
Time Frame: While on treatment with sulforaphane (less than or equal to 20 weeks.)
Measure: Number; unit: percentage of participants
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
percentage of participants | 90

5. Secondary Outcome: Incidence of Grade 3 or Higher Treatment Related Toxicity
Description: Toxicities will be graded based on the NIH Cancer Therapy Evaluation Program (CTEP) Common Toxicity Criteria of Adverse Events Version 4.0 (http://ctep.cancer.gov). All adverse events of any grade (for example, abnormal laboratory values, etc.) deemed clinically significant by the investigator will be recorded as a measure of the safety profile of sulforaphane
Time Frame: Continually through study and 14-30 days after last drug dose.
Measure: Number; unit: participants
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
participants | 0

6. Secondary Outcome: Half-life of Sulforaphane (SFN) in Blood
Time Frame: Day 1 of study treatment
Measure: Median (Full Range); unit: hours
Arm/Group | Sulforaphane
Number analyzed (Participants) | 20
hours | 2.2 [1.8 to 5.5]

7. Secondary Outcome: Half-life of SFN in Blood Among Patients With Glutathione-S-Transferase Mu 1 (GSTM1) Null Genotype
Time Frame: Day 1 of study treatment
Measure: Median (Full Range); unit: Hours
Arm/Group | Sulforaphane
Number analyzed (Participants) | 8
Hours | 2.6 [2.0 to 5.5]

8. Secondary Outcome: Half-life of SFN in Blood Among Patients With Glutathione-S-Transferase Mu 1 (GSTM1) Intact Genotype
Time Frame: Day 1 of study treatment
Measure: Median (Full Range); unit: hours
Arm/Group | Sulforaphane
Number analyzed (Participants) | 12
hours | 2.1 [1.8 to 2.9]

ADVERSE EVENTS:
Groups:
- Sulpforaphane: Sulforaphane given 200μmol (total daily) orally in four 50μmol capsules taken once daily from Week 1 Day 1 to Week 20 Day 7. On days when clinic visits are required patient must wait to take that day's dose until instructed to do so in clinic
Arm/Group | Sulpforaphane
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulpforaphane (N=20)
Bloating (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 7
Gatrointestinal pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes